CLINICAL TRIAL: NCT04175964
Title: Role of the Ketogenic Diet in Women With PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mazen Abdel Rasheed, Researcher, Principal Investigator, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ketogenic diet in PCOS
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet, Ketogenic; Metformin; Caloric Restriction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): PCO patients that will receive ketogenic diet only
  Interventions: Behavioral: ketogenic diet
- Group 2 (Experimental): PCO patients that will receive caloric diet with Metformin
  Interventions: Combination Product: caloric diet with Metformin
- Group 3 (Experimental): PCO patients that will receive caloric diet only
  Interventions: Behavioral: caloric diet

INTERVENTIONS:
Behavioral: ketogenic diet — The ketogenic diet will be designed according to the BMI for each participant by a consultant nutritionist. All participants will be prescribed this diet for 8 weeks.
  Arms: Group 1
Combination Product: caloric diet with Metformin — The caloric diet will be designed according to the BMI for each participant by a consultant nutritionist. All participants will be prescribed this diet with Metformin for 8 weeks.
  Arms: Group 2
Behavioral: caloric diet — The caloric diet will be designed according to the BMI for each participant by a consultant nutritionist. All participants will be prescribed this diet for 8 weeks.
  Arms: Group 3

SUMMARY:
For the fact of PCOS symptoms could be improved with weight loss and improving insulin resistance, the investigators will do this study to evaluate the role of the ketogenic diet in overweight and obese women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is one of the most common endocrinal abnormalities that affect females within the reproductive age, and are found in about 4% of women. PCOS is commonly associated with symptoms of increased testosterone such as irregular or absent menstrual cycle, increased body hair, and infertility. PCOS is also associated with other disorders such as obesity, insulin resistance, hyperinsulinemia, diabetes mellitus type 2, and dyslipidemia.

Until now, there is no known curative treatment for PCOS. However, anti-diabetic medications can improve many metabolic disorders such as insulin resistance, and increased levels of serum testosterone and total cholesterol. In addition, regulation of diet with exercise could improve the insulin sensitivity. Therefore, managements that aim to decrease the insulin level, improve the insulin resistance and decrease the body weight may be useful for improving symptoms of PCOS.

Ketogenic diets are characterized by a reduction in carbohydrates (usually to less than 50 g/day) and a relative increase in the proportions of protein and fat. People following the keto diet gain 75% of their calories from fat, 20% from protein, and 5% from carbohydrates. Previous studies have revealed that the ketogenic diet of low carbohydrate could decrease the body weight and improve the insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 16-35 years.
2. BMI ≥ 27.
3. Normal Renal Function.
4. Rotterdam criteria for the diagnosis of polycystic ovary syndrome:

   * Oligo/anovulation
   * Hyperandrogenism
   * Polycystic ovaries on ultrasound.

Exclusion Criteria:

1. Age <16 or >35 years.
2. BMI < 27.
3. Pregnancy.
4. Major medical disorders or other concurrent medical illnesses e.g. DM, other causes of androgen excess and hypercholesteremia
5. Current or previous use of hormonal, anti-diabetic or anti-obesity drugs, or other drugs that affect hormone levels, carbohydrate metabolism or appetite.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Role of the ketogenic diet in restoring normal ovulation that will be assessed by serial transvaginal ultrasound. | 8 weeks
  To evaluate the role of the ketogenic diet in overweight and obese women with PCOS regarding ovulation that will be assessed by serial transvaginal ultrasound.
comparison between ketogenic diet, caloric diet and caloric diet with Metformin regarding ovulation that will be assessed by serial transvaginal ultrasound. | 8 weeks
  comparison between ketogenic diet, caloric diet and caloric diet with Metformin regarding ovulation that will be assessed by serial transvaginal ultrasound.

SECONDARY OUTCOMES:
Role of the ketogenic diet in the affection of testosterone level | 8 weeks
  To evaluate the role of the ketogenic diet in the affection of testosterone level in overweight and obese women with PCOS
comparison between ketogenic diet, caloric diet and caloric diet with Metformin regarding testosterone level | 8 weeks
  comparison between ketogenic diet, caloric diet and caloric diet with Metformin regarding testosterone level

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abbassy, MD, Study Director — National Research Centre, Egypt

REFERENCES:
- [Background] Mavropoulos JC, Yancy WS, Hepburn J, Westman EC. The effects of a low-carbohydrate, ketogenic diet on the polycystic ovary syndrome: a pilot study. Nutr Metab (Lond). 2005 Dec 16;2:35. doi: 10.1186/1743-7075-2-35. PMID 16359551
- [Background] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291
- [Background] Moran LJ, Noakes M, Clifton PM, Tomlinson L, Galletly C, Norman RJ. Dietary composition in restoring reproductive and metabolic physiology in overweight women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2003 Feb;88(2):812-9. doi: 10.1210/jc.2002-020815. PMID 12574218